CLINICAL TRIAL: NCT00868283
Title: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Evaluate the Safety and Efficacy of Cerebrolysin in Patients With Acute Ischemic Stroke
Brief Title: The Safety and Efficacy of Cerebrolysin in Patients With Acute Ischemic Stroke
Acronym: CASTA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ever Neuro Pharma GmbH (Industry)
Collaborators: Excel PharmaStudies, Inc. (Industry); idv Datenanalyse und Versuchsplanung (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EBE-CN-050823
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — cerebrolysin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cerebrolysin (Experimental)
  Interventions: Drug: Cerebrolysin
- 0.9% Saline Solution (Placebo Comparator)
  Interventions: Drug: 0.9% Saline Solution

INTERVENTIONS:
Drug: Cerebrolysin — 30 ml study drug will be given once daily by intravenous infusion for 10 consecutive days.
  Arms: Cerebrolysin
Drug: 0.9% Saline Solution — 30 ml will be given once daily by intravenous infusion for 10 consecutive days.
  Other Names: NaCl
  Arms: 0.9% Saline Solution

SUMMARY:
The study investigated the clinical efficacy and safety of a 10-day course of therapy with daily intravenous administration of 30mL Cerebrolysin based on a comparison with Placebo in patients with acute ischemic stroke. 1070 patients were randomized in this trial in 2 parallel groups, one receiving Cerebrolysin, the control group receiving Placebo. Study drug will be given once daily by intravenous infusion for 10 consecutive days. Acetylsalicylic acid will be given orally, once daily throughout the study duration of 90 days as basic treatment. The clinical observation period for each patient will be 3 months and will include six clinical evaluation visits at Baseline (day 1) and on study days 2, 5, 10, 30 and 90.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years
* Focal neurological deficit
* Clinical diagnosis of acute hemispheric ischemic stroke
* CT or MRI results compatible with clinical diagnosis of acute hemispheric stroke
* NIH Stroke Scale Score between 6 and 22, both inclusive
* Functionally independent prior to stroke with a pre-stroke Rankin Score of 0 or 1
* Randomization and first treatment with the trial medication within 12h after stroke onset
* Informed consent given by the patient and/or the patient's legally acceptable representative

Exclusion Criteria:

* Evidence on CT/MRI of acute or chronic intracerebral hemorrhage, SAH, AVM, cerebral aneurysm, or neoplasm
* Signs of herniation, increased intracranial pressure or likely etiology other than brain ischemia at baseline CT scan
* Patients with a substantial decrease of consciousness or alertness at the time of randomization, defined as score of 2 or more one of the NIH Stroke Scale questions 1a.
* Neurological signs and symptoms that improve rapidly during screening and are likely to resolve completely within 24h
* Severe coexisting systemic disease that significantly limits life expectancy
* Systolic blood pressure over 220 mmHg or diastolic blood pressure over 120 mmHg on repeated measurement (interval of 30 min) prior to study entry
* Severe congestive heart failure or presentation with acute myocardial infarction at study entry
* Epilepsy or epileptic seizures at onset of stroke
* Pre-existing disorders or conditions that would impair interpretation of neurological assessment (eg. severe dementia, severe psychiatric illnesses, etc).
* Concomitant treatment with other neuroprotective or nootropic drugs (e.g. piracetam, citicoline, investigational neuroprotective substances)
* Patients which cannot tolerate or have contraindication to aspirin or Cerebrolysin treatment
* Concomitant treatment with substances that have a dilative effect on blood vessels like naftidrofuryl, cinnarizine, flunarizine or nimodipine
* Pregnancy and lactation period; for women with child-bearing potential a negative pregnancy test is required
* Participation in a clinical trial with an investigational drug in the past 4 weeks

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1071 (Actual)
Dates: Start 2006-09; Primary Completion 2010-10 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale | 90 days after start of treatment
Barthel Index | 90 days after start of treatment
NIH Stroke Scale | 90 days after start of treatment

SECONDARY OUTCOMES:
SF-12 | 90 days after start of treatment
Overall mortality | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Novak, PhD, Study Director — EVER Neuro Pharma; Zhen Hong, MD, Principal Investigator — Huashan Hospital, affiliated Fudan University
Locations (49):
- China (45):
  - Mudanjiang 1st people Hospital, Mudanjiang, Heilongjiang
  - Mudanjiang 2nd people Hospital, Mudanjiang, Heilongjiang
  - Anhui Shengli Hospital, Anhui
  - Anshan hospital, Anshan
  - Baotou Center Hospital, Baotou
  - Third hospital, affiliated Neimenggu Medical University (Bao Gang hospital), Baotou
  - Beijing PLA General Hospital, Beijing
  - First hospital, affiliated Peking University, Beijing
  - Friendship Hospital, affiliated Capital Medical University, Beijing
  - Peking Anzhen Hospital, Beijing
  - Sino-Japanese Friendship Hospital, Beijing
  - First hospital, affiliated Bethune Medical University, Changchun
  - Second Hospital Affiliated Bethune Medical University, Changchun
  - Xiangya Hospital, affiliated Hunan Medical University, Changsha
  - Chengdu 2nd People's Hospital, Chengdu
  - First Hospital, affiliated Huaxi Medical University, Chengdu
  - Sichuan Province People's Hospital, Chengdu
  - Second Hospital, affiliated Chongqing Med. University, Chongqing
  - Dalian Center Hospital, Dalian
  - Dalian third people Hospital, Dalian
  - Second Hospital, affiliated Wenzhou Med. University, Dalian
  - First hospital, affiliated Fujian Medical University, Fuzhou
  - FuJian Shengli Hospital, Fuzhou
  - First Hospital, affiliated Shantou Medical University, Guandong
  - Guangzhou 2nd People's Hospital, Guangzhou
  - Guangzhou red cross hospital, Guangzhou
  - First Hospital, affiliated Medical college Zhejing University, Hangzhou
  - The 4st Hospital affiliated Harbin Medical University, Harbin
  - Second Hospital, affiliated Kunming Med. University, Kunming
  - Yinchuan People's Hospital, Mudanjiang
  - Nanjing PLA General Hospital, Nanjing
  - Zhongda Hospital, Nanjing
  - First Hospital, affiliated Qingdao Medical University, Qingdao
  - Huashan Hospital, affiliated Fudan University, Shanghai
  - Renji Hospital, affiliated Second Medical University, Shanghai
  - Ruijin Hospital, affiliated Jiaotong University, Shanghai
  - Shanghai 6th People's Hospital, Shanghai
  - Xinhua hospital of Shanghai Jiaotong University School of Medicine, Shanghai
  - Zhongshan Hospital, affiliated Fudan University, Shanghai
  - Hebei Province People's Hospital, Shijiazhuang
  - Tianjin First Medical Center, Tianjin
  - Tianjin Union Medicine Centre, Tianjin
  - Union Hospital, affiliated Huazhong science and technology University, Wuhan
  - First hospital, affiliated NingXia Mededical University, Yinchuan
  - First hospital, affiliated Henan Medical University, Zhengzhou
- Chinese University of Hong Kong, Hong Kong, Hong Kong
- South Korea (3):
  - Asan medical center, Seoul
  - East-west neo medical center, Seoul
  - Kyung-hee University Hospital, Seoul

REFERENCES:
- [Background] Hong Z, Moessler H, Bornstein N, Brainin M, Heiss WD; CASTA-Investigators. A double-blind, placebo-controlled, randomized trial to evaluate the safety and efficacy of Cerebrolysin in patients with acute ischaemic stroke in Asia--CASTA. Int J Stroke. 2009 Oct;4(5):406-12. doi: 10.1111/j.1747-4949.2009.00340.x. PMID 19765131
- [Result] Heiss WD, Brainin M, Bornstein NM, Tuomilehto J, Hong Z; Cerebrolysin Acute Stroke Treatment in Asia (CASTA) Investigators. Cerebrolysin in patients with acute ischemic stroke in Asia: results of a double-blind, placebo-controlled randomized trial. Stroke. 2012 Mar;43(3):630-6. doi: 10.1161/STROKEAHA.111.628537. Epub 2012 Jan 26. PMID 22282884
- [Result] Bornstein NM, Guekht A, Vester J, Heiss WD, Gusev E, Homberg V, Rahlfs VW, Bajenaru O, Popescu BO, Muresanu D. Safety and efficacy of Cerebrolysin in early post-stroke recovery: a meta-analysis of nine randomized clinical trials. Neurol Sci. 2018 Apr;39(4):629-640. doi: 10.1007/s10072-017-3214-0. Epub 2017 Dec 16. PMID 29248999
- See also: Results publication — http://www.ahajournals.org/doi/10.1161/STROKEAHA.111.628537?url_ver=Z39.88-2003&rfr_id=ori:rid:crossref.org&rfr_dat=cr_pub%20%200pubmed
- See also: Meta analytic results — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC5884916/